CLINICAL TRIAL: NCT05381701
Title: Evaluation Of Peroperative Atelectasis In Minimal, Low And Medium Flow Anesthesia By Lung Ultrasound Score
Brief Title: Effects of Different Flow Anesthesia on Atelectasis
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Tugce Ozturk, Anesthesiologist, Zonguldak Bulent Ecevit University
Other Study IDs: 2020/25-6
Record Dates: First submitted 2022-04-21; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Atelectasis; Due to Anesthesia; General Anesthesia; Low- Flow Anesthesia; Minimal Flow Anesthesia
Keywords: Lung Ultrasound Score; Minimal Flow Anesthesia; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Minimal Flow Anesthesia (0.25L/dk oxygen, 0,25 L/min air)
  Interventions: Procedure: Lung Ultrasound Score
- Group II: Low Flow Anesthesia (0.5L/dk oxygen, 0,5 L/min air)
  Interventions: Procedure: Lung Ultrasound Score
- Group III: Medium Flow Anesthesia (1L/dk oxygen, 1 L/min air
  Interventions: Procedure: Lung Ultrasound Score

INTERVENTIONS:
Procedure: Lung Ultrasound Score — Measuring the atelectasis area by ultrasound guidance from 12 different regions of the lung

SUMMARY:
Evaluation of atelectasis that may be caused by different flow rate anesthesia applications during the operation with lung ultrasound score.

ELIGIBILITY:
Inclusion Criteria:

* operation time 2-5 hours
* elective septoplasty and rhinoplasty
* ASA I-II

Exclusion Criteria:

* morbid obesity
* malignant hyperthermia
* opioid sensitivity
* alcohol or drug addiction
* congestive heart failure
* chronic obstructive pulmonary disease
* coronary artery disease
* anemia
* liver and kidney diseases
* pregnancy
* breast-feeding
* history of allergy to drugs used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I-II septoplasty and rhinoplasty patients aged 18-65 years
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
assessment of lung ultrasound score | Change from Baseline and 30 minute after emergence
  Effect of different flow anesthesia on lung ultrasound score

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Faculty of Medicine, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes